CLINICAL TRIAL: NCT06951048
Title: The Effects of Lower Extremity Neural Mobilization Techniques on Muscle Strength and Performance in Healthy Individuals
Brief Title: The Role of Lower Limb Neural Mobilization in Improving Balance and Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Selim Mahmut GÜNAY, Doctor of Physical Therapy, Uludag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2025/4-1
Record Dates: First submitted 2025-04-22; First posted 2025-04-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Healty Volunteers; Sedantary; Young; Female
Keywords: Neural Mobilisation; Performance; Balance; Reactive agility
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Neural Mobilization) (Experimental): This group will follow a neural mobilization protocol targeting the sciatic, femoral, and tibial nerves. Neural exercises will be applied using specific techniques to facilitate nerve sliding along its anatomical path. Each nerve mobilization will be performed in 4 sets of 10 repetitions, three times a week (non-consecutive days).
  Interventions: Other: Group I (Neural Mobilization)
- Group II (Neural Mobilization + Dynamic Stretching) (Active Comparator): This group will perform the same neural mobilization protocol as Group I, in addition to dynamic stretching exercises targeting the lower extremities. The dynamic stretching program includes active straight leg raises (SLR), vertical jumps, and 10-meter sprints, performed in 3 sets of 10 repetitions for each exercise.
  Interventions: Other: Group II (Neural Mobilization + Dynamic Stretching)
- Group III (Dynamic Stretching Only) (Active Comparator): This group will follow a dynamic stretching protocol consisting of the same SLR, vertical jump, and 10-meter sprint exercises, performed in 3 sets of 10 repetitions.
  Interventions: Other: Group III (Dynamic Stretching Only)

INTERVENTIONS:
Other: Group I (Neural Mobilization) — Participants will undergo a neural mobilization program targeting the sciatic, femoral, and tibial nerves. Exercises are designed to promote nerve sliding through specific movement patterns and are performed bilaterally. Each nerve mobilization is applied in 4 sets of 10 repetitions, three times per week on non-consecutive days, with 30-second rest intervals.
  Sciatic nerve: Performed in side-lying; ankle dorsiflexion with neck extension followed by dorsiflexion release and neck flexion.
  Femoral nerve: In side-lying; simultaneous movements of the hip, knee, and neck in flexion and extension.
  Tibial nerve: In supine; coordinated ankle, toe, and cervical spine movements with controlled hip/knee positioning.
  Arms: Group I (Neural Mobilization)
Other: Group II (Neural Mobilization + Dynamic Stretching) — Participants in this group will engage in the same neural mobilization protocol applied in Group I, combined with a structured dynamic stretching program targeting lower extremity flexibility and neuromuscular performance. The dynamic exercises include active straight leg raises (SLR), vertical jumps, and 10-meter sprints. Each activity will be performed in three sets of ten repetitions, aiming to enhance muscular activation, mobility, and functional readiness.
  Arms: Group II (Neural Mobilization + Dynamic Stretching)
Other: Group III (Dynamic Stretching Only) — This group will engage exclusively in a dynamic stretching protocol comprising active straight leg raises (SLR), vertical jump exercises, and 10-meter sprint drills. Each exercise will be performed in three sets of ten repetitions, focusing on enhancing lower extremity mobility, muscle activation, and functional movement capacity without any neural mobilization intervention.
  Arms: Group III (Dynamic Stretching Only)

SUMMARY:
Neural mobilization (NM) is a technique used to enhance the mobility of peripheral nerves relative to surrounding tissues, aiming to reduce physiological tension and improve movement quality. While its effects are well-documented in clinical populations, recent studies have explored its use in healthy individuals to improve flexibility, balance, and functional performance. Evidence supports its positive impact on hamstring flexibility; however, findings on balance and performance remain inconclusive. This study aims to examine the effects of lower extremity NM techniques on balance, flexibility, and functional performance in healthy individuals, addressing current gaps in the literature.

DETAILED DESCRIPTION:
Neural Mobilization (NM) is a therapeutic approach based on the movement of neural structures, applied either manually or through exercise. Neural tissue is mobilized relative to adjacent structures to reduce symptoms through mechanisms that may be mechanical or neurophysiological. The nervous system separates itself from surrounding tissues by considering its own mobility and the relationship with adjacent structures. NM can be applied through various stretching and mobilization maneuvers to either facilitate movement or maximize the sliding (gliding) of peripheral nerves relative to adjacent tissues.

Studies on both humans and animals have reported that NM reduces intraneural edema, improves intraneural fluid distribution, decreases thermal and mechanical hyperalgesia, and reverses increased immune responses. Although NM is commonly used to improve the functionality of neural structures and alleviate symptoms associated with disease, recent research has explored its application in asymptomatic individuals to influence flexibility and performance parameters and to prevent injuries.

Nunes et al. investigated changes in functional performance and balance parameters by applying lower extremity nerve mobilization to asymptomatic individuals. Their study concluded that a single session of NM (including both stretching and mobilization) applied to the sciatic, tibial, and femoral nerves in healthy subjects resulted in no significant changes in performance, suggesting that the dosage and duration of NM may influence the outcomes.

In their study examining the acute effects of neural gliding exercises on athletic performance in healthy individuals, Waldhelm et al. found that bilateral sciatic nerve gliding exercises did not outperform a dynamic stretching protocol in terms of performance. However, they reported a greater improvement in hamstring flexibility. Based on these findings, they suggested that incorporating NM into warm-up routines may help prevent injuries. Similarly, Sharma et al. stated that adding neural stretching or mobilization to static stretching contributed more to hamstring flexibility than static stretching alone, although no dynamic performance assessment was included in the study.

Another study investigated the effects of neurodynamic glide techniques on hamstring flexibility in healthy male football players aged. The results showed that the neurodynamic intervention group experienced significant improvements in hamstring flexibility one week later compared to the control group.

D'souza et al. evaluated the short-term effects of different neural mobilization techniques on hamstring flexibility in recreational football players. While both the neural stretching and neural mobilization groups showed significant improvements, there was no significant difference between the groups in terms of sit-and-reach and active knee extension test results.

Ferrera et al. investigated the acute effects of neural gliding and neural tensioning exercises on static postural control and jumping performance in football players. Both techniques resulted in significant improvements in measured parameters, though no significant differences were observed between the techniques. The positive effects were reported to last for approximately 30 minutes.

Although literature suggests that NM techniques contribute to flexibility in asymptomatic individuals, their effects on functional performance, balance, and posture remain controversial. Furthermore, the limited number of studies conducted on healthy populations and methodological variations in existing research create uncertainty regarding the efficacy of NM techniques. Therefore, there is a need for studies that examine the effects of application dosage and duration and contribute to the understanding of NM.

The aim of this study is to investigate the effects of lower extremity neural mobilization techniques on balance, flexibility, and functional performance in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Providing written informed consent to voluntarily participate in the study
* Being a female individual aged between 18 and 30 years
* Having no medical conditions that contraindicate participation in physical exercise

Exclusion Criteria:

* Presence of structural spinal deformities such as scoliosis
* History of lumbar or lower extremity surgery within the past 12 months
* Experience of localized pain in the lumbar or lower extremity regions within the past 3 months
* Diagnosis of any neurodegenerative or neuromuscular disorders
* Presence of any medical condition that may hinder or contraindicate safe participation in exercise interventions

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Reactive Agility Test | Baseline and at Week 2
  Y-shaped course will be set up using three cones spaced 2 meters apart. Participants start by sprinting from the starting line; at the middle cone, a test administrator will randomly direct them to run left or right toward the finish line. Time will be recorded from the start to finish, and the best of three trials will be used for analysis.
Y Balance Test | Baseline and at Week 2
  This test assesses balance and stability. Participants will reach in three directions: anterior, 135° posteromedial, and 135° posterolateral using a prepared setup. After six practice attempts per direction, three test trials will be recorded, and the best score will be used. Lower limb length will be measured from the anterior superior iliac spine to the medial malleolus.
Active Straight Leg Raise Test | Baseline and at Week 2
  Used to assess hamstring flexibility. The test leg is lifted straight (without knee flexion) three times, and the highest angle of hip flexion measured with a goniometer will be recorded.
Muscle Strength | Baseline and at Week 2
  Isometric strength of the lower extremity will be measured using the Lafayette Manual Muscle Testing System Model-01165 (Lafayette Instrument Company, Lafayette IN, USA). Maximum isometric contraction will be measured in both knee flexion and extension with participants seated at 90° hip and knee flexion. Each contraction will last 5 seconds, repeated three times, and the average value will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Uludag University, Bursa, Nilüfer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding participant privacy and limitations in the informed consent obtained from participants

REFERENCES:
- [Background] Castellote-Caballero Y, Valenza MC, Martin-Martin L, Cabrera-Martos I, Puentedura EJ, Fernandez-de-Las-Penas C. Effects of a neurodynamic sliding technique on hamstring flexibility in healthy male soccer players. A pilot study. Phys Ther Sport. 2013 Aug;14(3):156-62. doi: 10.1016/j.ptsp.2012.07.004. Epub 2012 Nov 8. PMID 23142014
- [Background] Waldhelm A, Gacek M, Davis H, Saia C, Kirby B. ACUTE EFFECTS OF NEURAL GLIDING ON ATHLETIC PERFORMANCE. Int J Sports Phys Ther. 2019 Jul;14(4):603-612. PMID 31440411
- [Background] Ferreira J, Bebiano A, Raro D, Martins J, Silva AG. Comparative Effects of Tensioning and Sliding Neural Mobilization on Static Postural Control and Lower Limb Hop Testing in Football Players. J Sport Rehabil. 2019 Nov 1;28(8):840-846. doi: 10.1123/jsr.2017-0374. PMID 30222495
- [Background] Heredia Macias C, Paredes Hernandez V, Fernandez Seguin LM. A systematic review of the efficacy of neural mobilisation in sport: A tool for the neural tension assessment. J Bodyw Mov Ther. 2024 Oct;40:1409-1416. doi: 10.1016/j.jbmt.2023.04.034. Epub 2023 Apr 17. PMID 39593463
- [Derived] Gunay SM, Erturk E. Effects of lower limb neural mobilisation on reactive agility, balance, and physical performance: a randomised controlled trial. BMC Sports Sci Med Rehabil. 2025 Dec 10;18(1):1. doi: 10.1186/s13102-025-01461-3. PMID 41372947
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39593463/